CLINICAL TRIAL: NCT02863289
Title: Proximal Humerus Fractures in Children: The Outcomes of Conservative Management
Brief Title: The Outcomes of Proximal Humerus Fractures in Children
Status: Completed | Type: Observational
Sponsor: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Ben Clift, Mr. Ben Clift, NHS Tayside
Other Study IDs: 2016PB01
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-11

CONDITIONS: Humeral Fractures
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children with proximal humerus fractures: Children aged from 10 to 18-year-old in NHS Tayside whom sustained proximal humerus fractures during year 2008 to 2015.

SUMMARY:
To date, the clinical benefits and harms of surgical intervention in proximal humerus fractures in children remain debatable. The practical question raised by orthopaedic surgeons is: for children and adolescent, are the clinical and radiological outcomes after non-operative management as equivalent as after surgical management for proximal humerus fractures? The investigators' hypothesis is that due to the healing potential of the proximal humerus, the outcome from this fracture is usually excellent.

The investigators have applied for Caldicott approval to identify a cohort of eligible patient from NHS Tayside's radiography service. With the community health index (CHI) number, the investigators can review all shoulder X-rays performed in children and adolescents, aged from 10 to 18-year-old in NHS Tayside, from 2008 to 2015. The Caldicott approval also allowed the investigators to obtain clinical communication from the Clinical Portal (electronic summary healthcare records). The investigators will then conduct mail questionnaires, based on the Upper Extremities Functional Index (UEFI). The investigators will send out invitation letter with participation information and the UEFI questionnaires to the eligible patients; with return postages. If no response within 2 weeks, the investigators will send out 1 further reminder. If no further response, the patient will be excluded from the study.

DETAILED DESCRIPTION:
Proximal humerus fractures in children are relatively uncommon and most of them do not require surgical treatment due to the healing potential in children. The management of proximal humerus fractures in children subsequently underwent a major change with the introduction of surgical metal rod nailing. Despite that, the best criteria for choosing between these two treatment options are still not agreed upon. To date, the clinical benefits and harms of surgical intervention in proximal humerus fractures in children remain debatable. The investigators hypothesised that the outcomes of the non-operative management for proximal humerus fractures to remain excellent due to the healing ability of children. If good clinical results are achieved in our patient cohort, the investigators would like to send out the message that non-operative treatment for proximal humerus fractures in children should be recommended, even for those severely displaced fractures.

With Caldicott approval, the investigators can review the X-rays performed in children and adolescents, aged from 10 to 18-year-old in NHS Tayside, from 2008 to 2015. By using the Picture Archiving and Communication System (PACS), the investigators will be able to identify the cohort of patients who had proximal humerus fractures from the X-rays. The Caldicott approval also allowed the investigators to obtain clinical communication from Clinical Portal. The identified potential participants will be approached by the paediatric orthopaedic team. An invitation letter, a participant information sheet and questionnaire, based on UEFI will be sent to all potential participants by the care team via post. If no response within 2 weeks, the investigators will send out 1 further reminder. If no further response, the patient will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Within age limit
* Had proximal humerus fracture within study year
* Return questionnaire

Exclusion Criteria:

* No proximal humerus fractures
* Not return mail questionnaire

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged from 10 to 18-year-old in NHS Tayside who had proximal humerus fractures during year 2008 to 2015.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wei Lim, Principal Investigator — NHS Tayside

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 01/11/2016 to 01/03/2017 in Tayside.
Pre-assignment Details: All children who sustained proximal humerus fracture at age of 10 to 18 years old in Tayside.
Groups:
- Children With Proximal Humerus Fractures: Children aged from 10 to 18-year-old in NHS Tayside who sustained proximal humerus fractures during year 2008 to 2015.
Period: Overall Study
Arm/Group | Children With Proximal Humerus Fractures
Started | 118 (Study started on 01/11/2016, with 118 study participants.)
Completed | 35 (Study completed on 01/03/2017, 35 study participants have returned the questionnaire.)
Not Completed | 83

BASELINE CHARACTERISTICS:
Arm/Group | Children With Proximal Humerus Fractures
Number analyzed (Participants) | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 118
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 12 [10 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 62
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Indicated Status as Assessed by Mail Questionnaire Upper Extremities Functional Index (UEFI)
Description: Mail questionnaires based on the Upper Extremities Functional Index (UEFI) with return postages were sent out to the eligible cohort. UEFI range between 0 to 59, where the higher the UEFI, the better the functional outcomes.
Time Frame: From year 2008 to 2015
Measure: Count of Participants; unit: Participants
Arm/Group | Children With Proximal Humerus Fractures
Number analyzed (Participants) | 35
Participants
  Presence of Pain | 4
  Any difference between injured and non-injured arm | 4
  UEFI of 59 points | 24

2. Secondary Outcome: Number of Participants With Indicated Outcomes as Assessed by Radiological Parameters
Description: All shoulder X-rays performed in patients aged from 10 to 18-year-old and from 2008 to 2015 were reviewed. Radiological parameters, including degree of displacement and angulation; and any radiological residual deformities were recorded.
Time Frame: From year 2008 to 2015
Measure: Count of Participants; unit: Participants
Groups:
- Radiological Outcomes: The radiological parameters of all 118 study participants
Arm/Group | Radiological Outcomes
Number analyzed (Participants) | 118
Participants
  Surgical neck fracture | 91
  Presence of displacement | 56
  Presence of angulation | 84
  Residual angulation at follow up | 55
  Worsened angulation | 25

ADVERSE EVENTS:
Time Frame: 4 months.
Arm/Group | Children With Proximal Humerus Fractures
Serious Adverse Events (participants affected / at risk) | 0/118
Other Adverse Events (participants affected / at risk) | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes